CLINICAL TRIAL: NCT05211544
Title: The Effect of Physical Therapy Modalities and Kinesio Taping on Kinesiophobia and Thickness of the Quadriceps Muscle in Patients With Knee Osteoarthritis
Brief Title: The Effect of Physical Therapy Modalities and Kinesio Taping in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ayşe özdemirkan, medical doctor, Abant Izzet Baysal University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ao...1
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis; Knee Pain Chronic
Keywords: kinesio tape; kinesiophobia; therapeutic ultrasound; exercise; ultrasound
MeSH Terms: conditions — Osteoarthritis, Knee; Kinesiophobia; Motor Activity | interventions — Physical Therapy Modalities; Exercise

STUDY DESIGN:
Intervention Model Description: three group
  1. exercise group
  2. exercise and kinesiotape
  3. exercise and physical therapy modalities
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intervention group 1 (Active Comparator): 30 patient with osteoartritis will do knee strengthening exercise for half an hour a day,3 days a week. This exercise program will continue for 4 weeks. Also they will receive physical therapy modalities during two weeks for ten times. physical therapy modalities include hotpack, tens, ultrasound.
  Interventions: Other: physical therapy modalities and exercise
- intervention group 2 (Active Comparator): 30 patient with osteoartritis will do knee strengthening exercise for half an hour a day,3 days a week. This exercise program will continue for 4 weeks. Also they will receive kinesio tape for their knee three times a week for two week
  Interventions: Other: kinesio taping and exercise
- control group (Active Comparator): 30 patient with osteoartritis will do knee strengthening exercise for half an hour a day,3 days a week. This exercise program will continue for 4 weeks.
  Interventions: Other: exercise

INTERVENTIONS:
Other: physical therapy modalities and exercise — 30 patient with osteoartritis will do knee strengthening exercise for half an hour a day,3 days a week. This exercise program will continue for 4 weeks. Also they will receive physical therapy modalities during two weeks for ten times. physical therapy modalities include hotpack, tens, ultrasound.
  Arms: intervention group 1
Other: kinesio taping and exercise — 30 patient with osteoartritis will do knee strengthening exercise for half an hour a day,3 days a week. This exercise program will continue for 4 weeks. Also they will receive kinesio tape for their knee three times a week for two week
  Arms: intervention group 2
Other: exercise — 30 patient with osteoartritis will do knee strengthening exercise for half an hour a day,3 days a week. This exercise program will continue for 4 weeks.
  Arms: control group

SUMMARY:
Osteoarthritis (OA) is the most common degenerative joint disease with pathological structural and functional disorders all over the world. 27 million patients diagnosed with osteoarthritis in the USA alone.(1-2)

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common degenerative joint disease with pathological structural and functional disorders all over the world. 27 million patients diagnosed with osteoarthritis in the USA alone.(1-2) The primary risk factor for OA is age however ; It is a multifactorial disease, including injury and genetic mutations.(3-6) The knee is the most commonly involved joint in OA. In the United States, about 14 million people is presumed to have symptomatic knee osteoarthritis. Typical OA manifests as joint pain which is exacerbated by activity and relieved by rest. In advanced stage, pain at rest and at night and morning stiffness lasting no more than 20-30 minutes can be seen. (2) The diagnosis is based on a detailed anamnesis, a complete physical examination, and diagnostic imaging. Imaging findings include joint space narrowing, osteophytes, pseudocyst and subchondral sclerosis in the subchondral bone.(9) Pharmacological and non-pharmacological treatments are applied. Exercise, conventional physical therapy ( hotpack, therapeutic ultrasound, tens) and kinesioband are some of the non-pharmacological treatments.

ELIGIBILITY:
Inclusion Criteria:

over 50 ages Stage 2-3 osteoarthritis according to Kellgren Lawrence lectures

Exclusion Criteria:

Presence of acute infection The patient has a history of knee surgery Presence of rheumatological disease History of malignancy Major knee trauma Presence of crystal arthropathy Presence of acute trauma/fracture History of avascular necrosis The presence of contracture in the knee Using analgesic or anti-inflammatory drugs in the last 1 week Using oral or intramuscular corticosteroids in the last 3 months Intra-articular injection of the knee in the last 6 months Receiving physical therapy modalities from the knee area in the last 1 year Diseases such as dementia that may cause loss of cognitive functions

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-01-21 (Estimated); Primary Completion 2022-03-21 (Estimated); Study Completion 2022-04-21 (Estimated)

PRIMARY OUTCOMES:
tampa scala of kinesiophobia | four weeks
  It is developed to measure the fear of movement and reinjury. The scale will be measured at the beginning of the study and at the end of the fourth week, which corresponds to the end of the treatment
thickness of the quadriceps muscle | four weeks
  Muscle hypertrophy is expected with regular isometric and isotonic exercises. In order to investigate the muscle effect of the treatments, the thickness of the quadriceps muscle will be measured with an ultrasound device. Measurement will be made at the beginning of the study and at the end of the fourth week, which corresponds to the end of the treatment

SECONDARY OUTCOMES:
western ontario and mcmaster universities osteoarthritis index | four weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a widely used, to evaluate the condition of patients with osteoarthritis of the knee and hip, including pain, stiffness, and physical functioning of the joints. Measurement will be made at the beginning of the study and at the end of the fourth week, which corresponds to the end of the treatment
visual analog scale | four weeks
  The visual analog scale (VAS) is used to measure pain. The patient indicates where his/her condition is appropriate above a 100 mm line. For example, for pain, there is no pain at one end and very severe pain at the other end, and the patient marks his/her condition on this line. Measurement will be made at the beginning of the study and at the end of the fourth week, which corresponds to the end of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No